CLINICAL TRIAL: NCT02260284
Title: The Effect of Acupuncture in Treating Chronic Low-back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014LBP01
Record Dates: First submitted 2014-10-02; First posted 2014-10-09 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Ankylosing Spondylitis; Low Back Pain
MeSH Terms: conditions — Spondylitis, Ankylosing; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yaotong points acupuncture (Experimental): patients under the treatment of Yaotong ponts penetration mode
  Interventions: Other: Yaotong points acupuncture
- standardized acupuncture (Active Comparator): patients under the treatment of standardized acupuncture
  Interventions: Other: standardized acupuncture
- the usual care (Other): In the usual care group, participants received no study-related care-just the care, if any, that they and their physicians chose: mostly massage and physical therapy visits and continued use of medications (mostly nonsteroidal anti-inflammatory drugs (NSAIDS)).
  Interventions: Other: the usual care

INTERVENTIONS:
Other: Yaotong points acupuncture — Patients receive the treatments of Yaotong points penetration
  Arms: Yaotong points acupuncture
Other: the usual care — participants received no study-related care-just the care, if any, that they and their physicians chose: mostly massage and physical therapy visits and continued use of medications (mostly nonsteroidal anti-inflammatory drugs (NSAIDS))
  Arms: the usual care
Other: standardized acupuncture — Patients were given to the standardized acupuncture groups. This prescription included six acupuncture points that are commonly applied for the treatment of CLBP (Bladder 23-bilateral, Bladder 40-bilateral, and Kidney 3-bilateral) on the low back and lower leg.
  Arms: standardized acupuncture

SUMMARY:
The purpose of this study is to evaluate the efficiency of acupuncture in treating chronic low-back pain

DETAILED DESCRIPTION:
We want to know if the Yaotong points penetration or standardized acupuncture mode are more effective than medical care alone for CLBP; and if Yaotong points penetration is more effective than standardized acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* with CLBP
* without taking any other medication for the treatment of CLBP in at least 2 last weeks;
* aged from 18 to 50 years;
* without conflict to the written, informed consent signed prior to the enrollment.

Exclusion Criteria:

* pathological causes of chronic back pain (such as fractures, cancer, spinal stenosis and infections);
* complicated back problems (such as scoliologic >40° curvature, chronic spondylitis, sciatica, prior back surgery and other medicolegal issues);
* with contraindications for acupuncture (e.g., cardiac pacemakers, coagulation disfunctions, being in pregnancy, seizure disorder);
* conditions making treatment difficult (e.g., paralysis, psychoses);
* conditions that might confound treatment effects or interpretation of results (e.g., severe fibromyalgia, rheumatoid arthritis, concurrent care from other providers);
* previous acupuncture treatment for any condition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline on modified Roland-Morris Disability Questionnaire (RMDQ) at 24 weeks | at 0 week, 12 weeks, 24 weeks
  This wellvalidated questionnaire assesses pain on several dimensions including sensory pain, affective pain, and evaluative pain.

SECONDARY OUTCOMES:
Changes from baseline on Diagnosis and Curative Effect Standard for Syndrome of TCM for CLBP at 24 weeks | at 0 week, 12 weeks, 24 weeks
  It includes curing standard, referring to LBP had disappeared and no difficulty in movement was found; effective standard, referring to the pain was relieved but slight discomfort was found; and ineffective standard, referring to no symptom improvement was found.
Changes from baseline on short-form 36 health survey (SF-36) | at 0 week, 12 weeks, 24 weeks
  Physical and mental health component summary scores of the medical outcomes
Changes from baseline on Visual Analog Scale at 24 weeks | at 0 week, 12 weeks, 24 weeks
  This rating scale involved the selection of a point along a 10-cm line, which described pain intensity on a continuum from "no painat all" to "pain as bad as it could be." This scale has been found to be an excellent measure of self-reported pain

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Luo Y, Yang M, Liu T, Zhong X, Tang W, Guo M, Hu Y. Effect of hand-ear acupuncture on chronic low-back pain: a randomized controlled trial. J Tradit Chin Med. 2019 Aug;39(4):587-598. PMID 32186108